CLINICAL TRIAL: NCT02974738
Title: A Phase 1, Dose-Escalation and Expansion Trial of PT2977, a HIF-2α Inhibitor, in Patients With Advanced Solid Tumors
Brief Title: A Trial of Belzutifan (PT2977, MK-6482) Tablets In Patients With Advanced Solid Tumors (MK-6482-001)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Peloton Therapeutics, Inc., a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6482-001; PT2977-101 (Other: Pelaton Study ID); MK-6482-001 (Other: MSD)
Record Dates: First submitted 2016-11-23; First posted 2016-11-28 (Estimated); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Advanced Solid Tumors; Solid Tumor; Solid Carcinoma; Solid Tumor, Adult; ccRCC; RCC, Clear Cell Adenocarcinoma; RCC; Kidney Cancer; Clear Cell Renal Cell Carcinoma; Renal Cell Carcinoma, Metastatic; Renal Cell Carcinoma Recurrent; Renal Cell Carcinoma, Clear Cell Adenocarcinoma; Glioblastoma; Glioblastoma, Adult; GBM; Glioblastoma Multiforme
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms; Neoplasm Metastasis; Glioblastoma | interventions — belzutifan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Part 1A (Experimental): Drug: PART 1A: Belzutifan for the treatment of advanced solid tumors
  Belzutifan inhibits HIF-2α and is a novel approach to treatment of solid tumors.
  Interventions: Drug: Belzutifan
- Part 1B (Experimental): Drug: PART 1B: Belzutifan for the treatment of advanced ccRCC
  Belzutifan inhibits HIF-2α and is a novel approach to treatment of ccRCC.
  Interventions: Drug: Belzutifan
- Part 2 (Experimental): Drug: Part 2: Belzutifan for the treatment of other specified solid tumors
  Belzutifan inhibits HIF-2α and is a novel approach to treatment of specified solid tumors.
  Interventions: Drug: Belzutifan
- Part 2A (Experimental): Drug: Part 2A: Belzutifan for the treatment of patients with recurrent GBM who have been previously treated with radiation therapy and temozolomide
  Belzutifan inhibits HIF-2α and is a novel approach to treatment of specified solid tumors.
  Interventions: Drug: Belzutifan

INTERVENTIONS:
Drug: Belzutifan — Belzutifan is a highly selective small molecule that inhibits the function of the HIF-2α transcription factor. As a result, hypoxic signaling in cancer cells is impaired, blocking the transcription of several genes involved in oncogenesis
  Other Names: PT2977 Tablets, PT-2977, HIF-2α inhibitor, MK-6482; WELIREG™

SUMMARY:
The primary objective of this study is to identify the maximum tolerated dose (MTD) of belzutifan Tablets and/or the recommended Phase 2 dose (RP2D) of belzutifan Tablets in patients with advanced solid tumors

DETAILED DESCRIPTION:
Part 1A: This is a Phase 1, multiple-dose, dose-escalation trial of belzutifan Tablets, where patients with advanced solid tumors will be assigned to sequential dose cohorts. Patient safety will be monitored with frequent physical examinations, vital sign measurements, electrocardiograms (ECGs), and hematology and chemistry laboratory studies, and by recording all adverse events (AEs). Blood will be obtained for analysis of the concentration of belzutifan and to assess biomarkers.

Part 1B: Once the MTD and/or the RP2D is achieved, and expansion cohort of 50 patients with advanced clear cell renal cell carcinoma (ccRCC) will be enrolled.

Part 2: After determination of the MTD/RP2D, up to 25 patients with other specified solid tumors may be enrolled. Up to 3 different tumor types may be included in this part of the study.

Part 2A: A cohort of 25 patients with glioblastoma (GBM)

ELIGIBILITY:
Inclusion Criteria:

* Has a diagnosis of locally advanced or metastatic solid tumor
* Is of age ≥ 18 years
* Has a life expectancy of ≥ 6 months
* Has adequate organ function
* If a female patient, must not be pregnant or breastfeeding and not a woman of childbearing potential (WOCBP) OR a WOCBP who uses contraception or is abstinent from heterosexual intercourse during the study and for a minimum of 30 days after the last study drug administration, or if a male patient, must be abstinent from heterosexual intercourse OR agree to use contraception
* Able to swallow oral medications

Additional Inclusion Criteria for GBM cohort

* Must have histologically confirmed glioblastoma, IDH-wild type that is first recurrent following radiation therapy and temozolomide according to the Response Assessment in Neuro-Oncology (RANO) criteria
* Must have archival tumor tissue available from a previous surgery for glioblastoma
* Must have measurable (defined as at least 1 cm x 1 cm) contrast-enhancing lesion by MRI imaging within 21 days of starting treatment
* Must be able to undergo MRI of the brain with gadolinium. Patients must be maintained on a stable or decreasing dose of corticosteroid regimen (no increase for 5 days) prior to this baseline MRI
* Must have recovered from prior therapy to grade ≤1 severity (except for alopecia and lymphocytopenia) National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE)

Exclusion Criteria:

* Has a history of untreated brain metastasis or history of leptomeningeal disease or spinal cord compression
* Has failed to recover from the reversible effects of prior anticancer therapy (does not apply to GBM cohort)
* Has uncontrolled or poorly controlled hypertension
* Has malabsorption due to prior gastrointestinal (GI) surgery or GI disease
* Has had any major cardiovascular event within 6 months prior to study drug administration
* Has any other clinically significant cardiac, respiratory, or other medical or psychiatric condition that might interfere with participation in the trial or interfere with the interpretation of trial results
* Has had major surgery within 4 weeks before first study drug administration
* Has known HIV
* Has an active infection requiring systemic treatment
* Is participating in another therapeutic clinical trial

Additional Excusion Criteria for GBM cohort:

* Has received prior anti-VEGF therapy including bevacizumab (i.e. patients must be bevacizumab naïve)
* Is receiving enzyme-inducing anti-epileptic drugs (EIAED). Patients may be on non-enzyme inducing anti-epileptic drugs or not be taking any anti-epileptic drugs. Patients previously treated with EIAED may be enrolled if they have been off the EIAED for 10 days or more prior to the first dose of belzutifan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-12-07 (Actual); Primary Completion 2018-01-12 (Actual); Study Completion 2027-04-14 (Estimated)

PRIMARY OUTCOMES:
maximum tolerated dose (MTD) | 3 Weeks
  21-Day Dose Limiting Toxicity Observation Period per Dose Group

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Derived] Jonasch E, Bauer TM, Papadopoulos KP, Plimack ER, Merchan JR, McDermott DF, Dror Michaelson M, Appleman LJ, Roy A, Perini RF, Liu Y, Choueiri TK. Phase I LITESPARK-001 study of belzutifan for advanced solid tumors: Extended 41-month follow-up in the clear cell renal cell carcinoma cohort. Eur J Cancer. 2024 Jan;196:113434. doi: 10.1016/j.ejca.2023.113434. Epub 2023 Nov 15. PMID 38008031
- [Derived] Choueiri TK, Bauer TM, Papadopoulos KP, Plimack ER, Merchan JR, McDermott DF, Michaelson MD, Appleman LJ, Thamake S, Perini RF, Zojwalla NJ, Jonasch E. Inhibition of hypoxia-inducible factor-2alpha in renal cell carcinoma with belzutifan: a phase 1 trial and biomarker analysis. Nat Med. 2021 May;27(5):802-805. doi: 10.1038/s41591-021-01324-7. Epub 2021 Apr 22. PMID 33888901
- See also: Merck Oncology Clinical Trials Information — http://merckoncologyclinicaltrials.com